CLINICAL TRIAL: NCT04300192
Title: Immune Response to Pertussis After Vaccination With a Tdap-IPV Booster Vaccine in Children in the Republic of South Africa: Effect of Homologous and Heterologous Pertussis Vaccination Priming Background
Brief Title: Study to Evaluate the Immune Response After Booster Vaccination With Tdap-IPV Vaccine (Against Tetanus, Diphtheria, Pertussis and Poliomyelitis) in Children Who Received Different Pertussis Primary Vaccine Regimens in Republic of South Africa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TD500056; U1111-1223-5186 (Registry Identifier: ICTRP); TD500056 (Other: Sanofi Identifier); 2022-002452-40 (EudraCT Number)
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pertussis Immunisation; Diphtheria Immunisation; Tetanus Immunisation; Poliomyelitis Vaccine
MeSH Terms: interventions — Tetanus Toxoid; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1: Adacel Quadra vaccine (Experimental): Adacel Quadra single injection at Day 0 in participants who received 4 doses of whole-cell pertussis (wP) vaccine during the first 2 years of life
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine
- Group 2: Adacel Quadra vaccine (Experimental): Adacel Quadra single injection at Day 0 in participants who received 3 doses of wP followed by 1 dose of acellular pertussis (aP) vaccine during the first 2 years of life
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine
- Group 3: Adacel Quadra vaccine (Experimental): Adacel Quadra single injection at Day 0 in participants who received 2 doses of wP vaccine followed by 2 doses of aP vaccine during the first 2 years of life
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine
- Group 4: Adacel Quadra vaccine (Experimental): Adacel Quadra single injection at Day 0 in participants who received 1 dose of wP vaccine followed by 3 doses of aP vaccine during the first 2 years of life
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine
- Group 5: Adacel Quadra vaccine (Experimental): Adacel Quadra single injection at Day 0 in participants who received 4 doses of aP vaccine during the first 2 years of life
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine
- Group 6: Adacel Quadra vaccine (HIV positive) (Experimental): Adacel Quadra single injection at Day 0 in HIV + participants who received 4 doses of wP vaccine during the first 2 years of life
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine
- Group 7: Adacel Quadra vaccine (HIV positive) (Experimental): Adacel Quadra single injection at Day 0 in HIV + participants who received 4 doses of aP vaccine during the first 2 years of life
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine

INTERVENTIONS:
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Other Names: Adacel®-Polio, Adacel Quadra®

SUMMARY:
Primary Objectives :

* To describe the long-term humoral immune responses to pertussis, diphtheria, and tetanus after homologous and heterologous pertussis vaccine priming regimens
* To determine the effects of the priming regimen on humoral responses to booster vaccination with Tdap-IPV vaccine
* To describe the long-term cell-mediated immune responses to pertussis after homologous and heterologous pertussis vaccine priming regimens
* To determine the effects of the priming regimen on cell-mediated immune response to booster vaccination with Tdap-IPV vaccine

Secondary Objective:

To describe the safety profile of Tdap-IPV vaccine in each group

DETAILED DESCRIPTION:
Study duration per participant will be approximately 30 days including: 1 day of screening and vaccination, a phone call and a safety follow-up/end of study visit, at Day 8 and Day 30 after vaccine administration, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Born in 2007 to 2011 in the RSA
* Received primary pertussis vaccination and the toddler booster in the RSA
* Assent form has been signed and dated by the participant, and informed consent form (ICF) has been signed and dated by the parent(s) or another legal guardian and by an independent witness, if required by local regulations
* Participants and parent/legal guardian are able to attend all scheduled visits and to comply with all trial procedures
* Valid clinical record of primary vaccination with DTaP/DTwP vaccines immunization history from 2007 through 2011, either by hand-held (Road-to-Health Card) or immunization clinical records
* For Groups 6 and 7: children infected with perinatally acquired HIV infection currently under care who received either an all wP or all aP priming regimen
* For Groups 6 and 7: be on highly active antiretroviral therapy (HAART) therapy and have known CD4 cell counts > 200 cells/µL

Exclusion Criteria:

* Participation in the 4 weeks preceding the vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following the trial vaccination except for influenza
* Receipt of additional pertussis vaccination doses inconsistent with pertussis vaccination schedule in the RSA
* Previous confirmed diagnosis of pertussis disease
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* For Groups 1 to 5: known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known thrombocytopenia, as reported by the parent/ legal guardian or suspected thrombocytopenia contraindicating intramuscular vaccination in the Investigator's opinion
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Participants with progressive neurological disorder, uncontrolled epilepsy, or progressive encephalopathy except if a treatment regimen has been established and the condition has stabilized
* Encephalopathy within 7 days of a previous dose of pertussis-containing vaccine
* Had contraindication to receipt of Adacel Quadra vaccine at the time of vaccination as defined in the Adacel Quadra vaccine Republic of South Africa (RSA) label
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]). A prospective participants should not be included in the study until the condition has resolved or the febrile event has subsided (temporary contraindication)
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw Note: Potential participants receiving standard HIV treatments such as antiretrovirals and/or antibiotic prophylaxis can be enrolled in the study. Their routine medications should be documented in the CRB.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 273 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Concentrations (GMCs) of anti-pertussis total immunoglobulin G (IgG) | Day 0 (pre-vaccination) and Day 30 (post-vaccination)
  Total IgG anti-pertussis antibody concentrations against the following pertussis antigens: pertussis toxin (PT), filamentous hemagglutinin (FHA), pertactin (PRN), and fimbriae types 2 and 3 (FIM)
GMCs of anti-diphtheria IgG | Day 0 (pre-vaccination) and Day 30 (post-vaccination)
  Total IgG anti-diphtheria antibody concentrations
GMCs of anti-tetanus toxoid IgG | Day 0 (pre-vaccination) and Day 30 (post-vaccination
  Total IgG anti-tetanus antibody concentrations
GMCs of anti-pertussis total immunoglubulin A (IgA) and of anti-heat-killed B pertussis (HK Bp) IgA in cell-mediated immunity (CMI) subset only | Day 0 (pre-vaccination) and Day 30 (post-vaccination)
  Total IgA anti-pertussis antibody concentrations against the following pertussis antigens: PT, FHA, PRN, FIM types 2 and 3, and heat-killed B. pertussis (HK Bp)
Geometric Mean (GM) of anti-pertussis IgG subclasses and of anti-HK Bp IgG subclasses. | Day 0 (pre-vaccination) and Day 30 (post-vaccination)
  Anti-pertussis IgG subclasses (ie, IgG1, IgG2, IgG3, and IgG4) distribution against PT, FHA, PRN, FIM types 2 and 3, and HK Bp
GM of pertussis antigen-specific T cells | Day 0 (pre-vaccination) and Day 30 (post-vaccination)
  Absolute numbers (spot forming cells [SFC]/10e6 PBMCs) of pertussis antigen-specific (antigen pool and HK Bp) interferon (IFN)-ɣ, interleukin (IL)-17, IL-4 secreting cells

SECONDARY OUTCOMES:
Number of participants reporting immediate adverse events (AEs) | Within 30 minutes post-vaccination
  Medically relevant unsolicited systemic AEs, including those related to the product administered
Number of participants reporting solicited injection site reactions and systemic reactions | Within 7 days post-vaccination
  Adverse reactions prelisted in the (electronic) case report book (CRB) Injection site reactions: pain, erythema, swelling Systemic reactions: fever, headache, malaise, myalgia
Number of participants reporting unsolicited AEs | Within 30 days post-vaccination
  AEs other than solicited reactions
Number of participants reporting serious adverse events (SAEs) | Up to 37 days post-vaccination
  SAEs, including adverse event of special interest (AESIs)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- South Africa (3):
  - Investigational Site Number : 7100001, Cape Town
  - Investigational Site Number : 7100003, Johannesburg
  - Investigational Site Number : 7100002, Middelburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TD500056 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25353&tenant=MT_SNY_9011